CLINICAL TRIAL: NCT02476500
Title: Prospective Case-control Study to Assess the Construct Validity of a Large Loop Excision of the Transformation Zone (LLETZ) Training Model
Brief Title: Construct Validity of a Large Loop Excision of the Transformation Zone (LLETZ) Training Model
Acronym: LLETZ-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Clemens Tempfer, Prof. Clemens Tempfer, MD, Ruhr University of Bochum
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LLETZ-1
Record Dates: First submitted 2015-05-03; First posted 2015-06-19 (Estimated); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Cervical Dysplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experts (Active Comparator): Surgically experienced gynecologists with a personal history of at least 30 LLETZ procedures will undergo a Video Training and subsequently will perform LLETZ on a Training model. Their performance will be scored by using a 23-item OSATS scheme. The exact time Frame for the OSATS-assessment is within 1 hour after the Video Training.
  Interventions: Procedure: LLETZ on a training model
- Novices (Experimental): Medical students with no previous experience in gynecological surgery will undergo a Video Training and subsequently will perform LLETZ on a Training model. Their performance will be scored by using a 23-item OSATS scheme. The exact time Frame for the OSATS-assessment is within 1 hour after the Video Training.
  Interventions: Procedure: LLETZ on a training model

INTERVENTIONS:
Procedure: LLETZ on a training model — LLETZ is performed on a sausage-based training model using all surgical devices used in the original procedure

SUMMARY:
In a prospective case-control study, 140 medical students (,novices') and 10 Senior gynecologists (,experts') will perform a Large Loop Excision of the Transformation Zone (LLETZ) on a Training model afte having undergone a Video Training session. Their LLETZ-Performance will be assessed using an Objective Structured Assessment of Technical Skills (OSATS) protocol designed for judging the surgical proficiency when performing a LLETZ. Using metrical and non-metrical data points, construct validity of the LLETZ training model to distinguish between experts and novices will be assessed. Secondary endpoints are differences in OSATS scores within the group of novices based on gender and handyness, as well as satisfaction of the novices with the learning experience.

DETAILED DESCRIPTION:
In a prospective case-control study, 140 medical students (,novices') and 10 Senior gynecologists (,experts') will be included. All participants undergo a video training with demonstration of the LLETZ procedure on a training model using a sausage as previously described (Hefler et al. 2014). After the Video Training, the LLETZ procedure will be performed by the study probands and their performance will be assessed using an Objective Structured Assessment of Technical Skills (OSATS) protocol with 23 consecutive items. The exact time Frame for the assessment of the Primary outcome is within 1 hour after the Video Training. Using metrical and non-metrical items, the construct validity of the LLETZ training model to distinguish between experts and novices will be assessed. The study hypothesis is that the LLETZ Training model as used in this study has construct validity and is therefore a valid Instrument to discriminate between experts and novices. Secondary endpoints are differences in OSATS scores within the group of novices based on gender and handyness, as well as satisfaction of the novices with the learning experience.

ELIGIBILITY:
Inclusion Criteria:

* Medical Student
* no previous experience with the Training model
* no previous experience in gynecological surgery

Exclusion Criteria:

* language barrier
* unwillingness to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-05; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Construct validity | within 1 hour after the video training
  metric and non-metric OSATS points such as duration of surgery, cone volume resected, completeness of the cone

SECONDARY OUTCOMES:
Satisfaction | within 1 hour after the video training
  Subjects grade their satisfaction with the learning effect of the training model using a 5-step scale
Influence of gender on OSATS scores | within 1 hour after the video training
  OSATS scores will be compared according to the probands' gender
Influence of handyness on OSATS scores | within 1 hour after the video training
  OSATS scores will be compared according to the probands' handyness (right-handed versus left-handed)

CONTACTS AND LOCATIONS:
Overall Officials: Guenther A Rezniczek, PhD, Principal Investigator — Ruhr University Bochum
Locations (1):
- Dept. OBGYN Ruhr University Bochum, Herne, Germany

REFERENCES:
- [Result] Rezniczek GA, Severin S, Hilal Z, Dogan A, Krentel H, Buerkle B, Tempfer CB. Surgical performance of large loop excision of the transformation zone in a training model: A prospective cohort study. Medicine (Baltimore). 2017 Jun;96(23):e7026. doi: 10.1097/MD.0000000000007026. PMID 28591034